CLINICAL TRIAL: NCT06752109
Title: The Effect of Subtalar Joint Antipronation Taping on the Dynamic Knee Valgus in Female Volleyball Players with Low Medial Arch: a Double Blinded Randomized Controlled Trial
Brief Title: The Effect of Subtalar Joint Antipronation Taping on the Dynamic Knee Valgus in Female Volleyball Players with Low Medial Arch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Murat Akıncı, Msc, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTape01
Record Dates: First submitted 2024-12-17; First posted 2024-12-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Pes planus; ACL; Dynamic Tape
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Flatfoot | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Dynamic Tape
  Interventions: Other: Antipronation Taping
- Control (Sham Comparator): Sham Group
  Interventions: Other: Sham

INTERVENTIONS:
Other: Antipronation Taping — Before applying the tape, its length was measured by passing it over the areas on the foot where it would be applied. The tape was first attached to the medial side of the big toe, with tension in the direction of flexion and abduction of the toe. The ankle was then positioned in full plantar flexion. The tape was applied from the medial side of the foot towards the heel, wrapping around it, and then directed towards the sole. While the foot was in an inversion position at the navicular level, the tape was applied with maximum tension from medial to lateral and brought back to the sole. The remainder of the tape, with maximum tension, was applied from the sole to the dorsal side of the ankle, ending without tension at the proximal and lateral side of the leg. A second strip of tape, with maximum tension, was applied to support the medial longitudinal arch. The ends of the tape were placed over the malleoli without tension, aiming to reduce excessive pronation.
  Arms: Intervention
Other: Sham — In the sham taping application, the length of the tape was measured by passing it over the areas where it would be applied. The tape was applied to the medial side of the big toe, but without tension, simply placed. Then, the tape was directed towards the sole of the foot, passing over the heel. At the navicular level, the tape was applied from medial to lateral, returning to the sole without tension. A second strip of tape was applied to the sole without tension. The ends of the tape were placed over the malleoli without stretching. Since no tension was applied, this application was only placed and has a limited effect on reducing excessive pronation.
  Arms: Control

SUMMARY:
This study aims to investigate the biomechanical mechanisms of dynamic knee valgus and the impact of subtalar pronation, particularly due to decreased medial longitudinal arch, on knee injury risk, highlighting the importance of prevention and intervention strategies for athlete health.

DETAILED DESCRIPTION:
Dynamic knee valgus is an abnormal movement pattern of the lower extremity, formed by the combination of femoral adduction and internal rotation, tibial abduction and internal rotation, and subtalar pronation, and it is a significant risk factor for knee injuries. The foot and ankle represent the first link in the lower extremity kinetic chain, and a mechanical relationship between subtalar joint motion and tibial rotation triggers internal rotation of the tibia during weight-bearing. This is particularly more pronounced in female athletes, as increased foot pronation and medial longitudinal arch (MLA) drop contribute to dynamic knee valgus. Supporting the MLA has become increasingly important in injury prevention, as there is evidence in the literature showing that interventions to reduce foot pronation decrease dynamic knee valgus and help prevent patellofemoral pain and anterior cruciate ligament injuries.

The aim of this study is to investigate the effects of antipronation taping on dynamic knee valgus and knee flexion angle during functional jump tests in female volleyball players with MLA drop. Innovative taping materials, such as Dynamic Tape, when applied correctly, can support the MLA, reduce tibial rotation, and decrease abnormal movements. While there is existing evidence that MLA-supporting orthotics reduce such injury risks, no studies have specifically examined antipronation taping with Dynamic Tape applied to the subtalar joint. This study seeks to explore modifiable risk factors associated with common knee injuries in female athletes from a foot posture perspective and contribute to athlete health.

ELIGIBILITY:
Inclusion Criteria:

Actively playing volleyball for at least 5 years, A drop of 10 mm or more in the navicular drop test, A score of ≥ +4 according to the A foot posture index.

Exclusion Criteria:

A history of lower extremity injury within the last 3 months, A history of ankle and/or knee surgery, Having non-structural instability, A history of congenital or traumatic deformity in the lower extremity.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Single Leg Squat Test | Pre-taping and within 1 hour after taping
  In this test, athletes were instructed to perform a single-leg squat with their hands on their waist, maintaining balance for as long as possible, preferably for 5 seconds. Only trials that reached the required minimum flexion angle and maintained balance were considered valid. Three valid attempts were performed. During the tests, video recordings were made from both the front and the side. The footage was analyzed using the Microsoft OptoJump® Next program with a 2D analysis method to measure knee flexion and valgus angles.
Single Leg Landing Test | Pre-taping and within 1 hour after taping
  For this test, each athlete was asked to step off a 30 cm high box and extend the measurement leg forward to drop downward. The maximum knee valgus and flexion angles at the end of the drop were measured using two camera recordings, one from the front and one from the side.
  During the tests, video recordings were made from both the front and the side. The footage was analyzed using the Microsoft OptoJump® Next program with a 2D analysis method to measure knee flexion and valgus angles.
Vertical Drop Jump Test | Pre-taping and within 1 hour after taping
  In this test, athletes were instructed to stand with their feet shoulder-width apart on a 30 cm high box. They were then asked to jump into the square area in front of the box and immediately jump as far as possible using their arms for assistance. The test was completed once the athlete had made three successful jumps. The average of the three jumps was recorded.
  During the tests, video recordings were made from both the front and the side. The footage was analyzed using the Microsoft OptoJump® Next program with a 2D analysis method to measure knee flexion and valgus angles.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided